CLINICAL TRIAL: NCT06861270
Title: Estimation of Non-Reimbursable Direct Medical Costs, Direct Non-Medical Costs, and Indirect Costs for Patients With Duchenne Muscular Dystrophy in France
Brief Title: Estimation of Non-Reimbursable Costs for Patients With Duchenne Muscular Dystrophy in France
Acronym: CouDuMyo
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240695
Record Dates: First submitted 2024-09-25; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-07

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Duchenne muscular dystrophy (DMD) is a chronic neuromuscular disorder affecting approximately 150 to 200 newborns annually, predominantly males, and is characterized by progressive muscle atrophy and weakness due to a complete absence of dystrophin. DMD presents a severe phenotype, with life expectancy typically extending into the third decade. Data on healthcare utilization and associated costs for DMD patients, particularly within the French healthcare context, remain limited. The EPARDYS study aims to examine the care pathways of these patients using data from the Banque Nationale des Données Maladies Rares (BNDMR) and the Système National des Données de Santé (SNDS), enabling a detailed characterization of patient demographics, healthcare utilization patterns, and associated costs.

However, only direct costs eligible for reimbursement under the Affection Longue Durée (ALD 100%) scheme can be evaluated. Additional resources are consumed by DMD patients, particularly for medical care that falls outside the scope of reimbursement. Furthermore, the high level of dependency in these patients may lead to the need for home adaptations or other expenditures outside the healthcare domain but linked to the disease. Informal caregiving also plays a significant role.

These additional family-incurred costs must be considered. The CouDuMyo study will aim to estimate all relevant cost components from a societal perspective, considering both minors and adults, whether they attend school or work. The medico-social aspect of care, along with the collection of data on aids and benefits received, will offer insights into the nature of the support available to families in France. The knowledge gained regarding non-reimbursable, disease-related costs according to patient characteristics will provide a comprehensive view of the financial burden borne by patients and their caregivers. This assessment is particularly relevant in the context of emerging therapies, which may reduce these associated costs. The main objective will be to describe the resource utilization associated with DMD care that is not eligible for reimbursement, including direct medical costs not covered, medico-social expenses, direct non-medical costs, and indirect costs.

ELIGIBILITY:
The patients identified are those present in the BNDMR and with an up-to-date address for their follow-up centre.

Inclusion criteria

* Patients of any age with DMD diagnosed more than 6 months ago;
* Patient included in the BNDMR, not objecting to the collection of his or her data (see BNDMR 'Agreement to be contacted for a protocol') and alive at the time of his or her request to participate in the study.

Exclusion Criteria:

* Patient taking part in an interventional clinical study with changes to usual management (see BNDMR 'Patient taking part in a protocol');
* Patient and/or main carer objecting to the use of their data;
* Patient and/or main carer whose understanding of the French language does not allow them to complete the questionnaire.

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will focus on patients with Duchenne muscular dystrophy, whatever their age, and included in the BNDMR. This database brings together data on all patients treated in the rare disease expert centres approved by the DGOS, and shows a gross total of 2,028 patients with DMD on 1st March 2022.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Average annualised cost per patient/family. | 1 year
  The consumption of resources related to the care of patients with Duchenne muscular dystrophy (DMD) that are not eligible for reimbursement. This includes direct medical costs not covered by insurance, such as certain treatments, therapies, or medical devices that patients may require. Additionally, medico-social costs will be assessed, including services that support daily living and social integration, such as specialized transportation, caregiving, and educational support. Direct non-medical costs will also be evaluated, particularly those related to home modifications or equipment necessary for adapting the living environment to the patient's needs. Finally, the study will analyze indirect costs, which encompass the loss of productivity both for the patient and their caregivers, as well as the value of informal care provided by family members or other non-professional caregivers.

SECONDARY OUTCOMES:
Different types of costs identified for managing the disease | from disease identification to questionnaire's completion, up to 98 years
  All relevant expenses associated with the care of Duchenne muscular dystrophy (DMD) patients. The analysis will cover various categories of costs, including direct medical costs (both reimbursable and non-reimbursable), medico-social costs (such as home care or special education), direct non-medical costs (such as home adaptations or specialized equipment), and indirect costs (such as loss of productivity and informal caregiving)
Costs based on the severity of the disease | from disease identification to questionnaire's completion, up to 98 years
  How costs vary depending on the stage of disease progression. As DMD is a degenerative condition, the severity of the disease evolves over time, requiring different levels of care and resources at each stage. This analysis will examine how costs increase or change as the patient's functional abilities decline
Determinants of the identified costs | from disease identification to questionnaire's completion, up to 98 years
  The key factors that drive the costs of managing DMD. These determinants may include patient characteristics (such as age, disease duration, and comorbidities), socioeconomic factors (such as income, access to care, and geographic location), and the type of support or assistance available (such as public benefits, informal caregiving, and specialized services).

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Durand-Zaleski, Professor, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP Hôtel Dieu, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/70/NCT06861270/Prot_SAP_ICF_000.pdf